CLINICAL TRIAL: NCT02684292
Title: A Phase III, Randomized, Open-label, Clinical Trial to Compare Pembrolizumab With Brentuximab Vedotin in Subjects With Relapsed or Refractory Classical Hodgkin Lymphoma
Brief Title: Study of Pembrolizumab (MK-3475) vs. Brentuximab Vedotin in Participants With Relapsed or Refractory Classical Hodgkin Lymphoma (MK-3475-204/KEYNOTE-204)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-204; 163337 (Registry Identifier: JAPIC-CTI); MK-3475-204 (Other: MSD Protocol Number); KEYNOTE-204 (Other: MSD); 2022-500400-22-00 (Registry Identifier: EU CT); U1111-1275-8432 (Registry Identifier: UTN); 2015-005053-12 (EudraCT Number)
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Hodgkin Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg administered intravenously (IV) on Day 1 of each 3-week cycle for up to 35 cycles.
  Interventions: Biological: pembrolizumab
- Brentuximab vedotin (Active Comparator): Participants receive BV 1.8 mg/kg (maximum 180 mg per dose) IV on Day 1 of each 3-week cycle for up to 35 cycles.
  Interventions: Biological: brentuximab vedotin

INTERVENTIONS:
Biological: pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab
Biological: brentuximab vedotin — IV infusion
  Other Names: ADCETRIS®
  Arms: Brentuximab vedotin

SUMMARY:
The purpose of this study is to evaluate pembrolizumab (MK-3475) in the treatment of participants with relapsed or refractory Classical Hodgkin Lymphoma. Participants will be randomized to receive either pembrolizumab or brentuximab vedotin (BV) for up to 35 three-week cycles of treatment.

The primary hypotheses of this study are that treatment with pembrolizumab prolongs Progression-free Survival (PFS) and Overall Survival (OS) in participants with relapsed or refractory Classical Hodgkin Lymphoma compared to treatment with BV.

ELIGIBILITY:
Inclusion Criteria:

* Has relapsed (disease progression after most recent therapy) or refractory (failure to achieve Complete Response [CR] or Partial Response [PR] to most recent therapy) classical Hodgkin Lymphoma.
* Has responded (achieved a CR or PR) to BV or BV-containing regimens, if previously treated with BV.
* Has measurable disease defined as ≥1 lesion that can be accurately measured in ≥2 dimensions with spiral computed tomography (CT) scan or combined CT/positron emission tomography (PET) scan. Minimum measurement must be >15 mm in the longest diameter or >10 mm in the short axis.
* Is able to provide an evaluable core or excisional lymph node biopsy for biomarker analysis from an archival (>60 days) or newly obtained (within 60 days) biopsy at Screening (Visit 1).
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Has adequate organ function
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days (for participants receiving pembrolizumab) or 180 days (for participants receiving BV) after the last dose of study drug.
* Male participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 120 days (for participants receiving pembrolizumab) or 180 days (for participants receiving BV) after the last dose of study drug.

Exclusion Criteria:

* Has hypersensitivity to the active substance or to any of the excipients in BV or pembrolizumab.
* Is currently participating in or has participated in a study of an investigational agent and is currently receiving study therapy or has participated in a study of an investigational agent and has received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
* Has a diagnosis of immunosuppression or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has had a prior monoclonal antibody (mAb) within 4 weeks prior to first dose of study drug in the study or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy including investigational agents within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to a previously administered agent.
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. Note: Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of graft-versus-host disease (GVHD).
* Has a known additional malignancy that is progressing or requires active treatment in the last 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression by repeat imaging), clinically stable and without requirement of steroid treatment for ≥14 days prior to the first dose of study drug.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with the use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Has an active infection requiring intravenous systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days (for participants receiving pembrolizumab) or 180 days (for participants receiving BV) after the last dose of study drug.
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-PD-ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody (including ipilimumab) or OX-40 (Tumor necrosis factor receptor superfamily, member 4 [TNFRSF4]), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Has a known history of human immunodeficiency virus (HIV)
* Has active hepatitis B (HBV) or hepatitis C (HCV).
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis).
* Has received a live vaccine within 30 days prior to first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 40 months
Overall Survival (OS) | Up to approximately 40 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Kuruvilla J, Modi D, Santoro A, Paszkiewicz-Kozik E, Gasiorowski R, Johnson NA, Fogliatto LM, Goncalves I, de Oliveira J, Buccheri V, Perini GF, Goldschmidt N, Kriachok I, Sekiguchi N, Lin J, Yusuf R, Marinello P, Zinzani PL. Pembrolizumab in relapsed or refractory Hodgkin lymphoma: a post hoc analysis of KEYNOTE-204 by prior lines of therapy. Leuk Lymphoma. 2025 Sep;66(9):1710-1719. doi: 10.1080/10428194.2025.2502805. Epub 2025 Jun 23. PMID 40548833
- [Derived] Kuruvilla J, Ramchandren R, Santoro A, Paszkiewicz-Kozik E, Gasiorowski R, Johnson NA, Fogliatto LM, Goncalves I, de Oliveira JSR, Buccheri V, Perini GF, Goldschmidt N, Kriachok I, Dickinson M, Komarnicki M, McDonald A, Ozcan M, Sekiguchi N, Zhu Y, Nahar A, Marinello P, Zinzani PL; KEYNOTE-204 investigators. Pembrolizumab versus brentuximab vedotin in relapsed or refractory classical Hodgkin lymphoma (KEYNOTE-204): an interim analysis of a multicentre, randomised, open-label, phase 3 study. Lancet Oncol. 2021 Apr;22(4):512-524. doi: 10.1016/S1470-2045(21)00005-X. Epub 2021 Mar 12. PMID 33721562
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26185&tenant=MT_MSD_9011